CLINICAL TRIAL: NCT01014923
Title: Parent-based Intervention to Increase Safe Teen Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Blank Children's Hospital (Other)
Responsible Party: Corinne Peek-Asa, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE000947; CDC NCIPC R49 CE000947
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Motor Vehicle Occupant Injury; Teenaged Driver
Keywords: motor vehicle; accidents, traffic; prevention and control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Parents of new teen drivers receive guidebook to teach driving skills and safety behaviors; individual instruction on parent-child communication about driving; DVD demonstrating safe driving communication; and, 26-page booklet on driving goals and conversation topics
  Interventions: Behavioral: Teen driving intervention
- Control (No Intervention): Parents receive a Department of Transportation booklet on teen driving

INTERVENTIONS:
Behavioral: Teen driving intervention — Parents of new teen drivers receive guidebook to teach driving skills and safety behaviors; individual instruction on parent-child communication about driving; DVD demonstrating safe driving communication; and, 26-page booklet on driving goals and conversation topics
  Arms: Intervention

SUMMARY:
We hypothesize that this intervention will increase the quality and quantity of parental interaction on safety driving with newly-licensed teen drivers. 250 parent/teen dyads will be individually randomized into intervention and control groups. The intervention group will receive a tailored, in-person intervention with a trained member of the research team, with follow-up intervention phone calls each month for the 3-month intervention. The control group will be a "usual care" group who will receive driving safety materials available to all new drivers and their parents. Parents and teens will be followed to see if intervention parents meet the intervention's driving goals and to see if the parent and teens report improved driving skills and behaviors in the intervention compared with the control group.

DETAILED DESCRIPTION:
Drivers in their first six months of licensure have the highest crash rates of all drivers, leading to high rates of injury for themselves, their passengers, and those they hit. Parents play a critical role in the driving experience of their children. Policy approaches, such as Graduated Driver's Licensing Systems, and educational programs that encourage parents to define driving rules and restrictions have shown some success in reducing teen risky driving. However, methods to increase parental involvement in teaching driving skills and encouraging safe driving behaviors have not been widely tested. Such interventions can augment existing GDL systems by increasing parental knowledge and involvement in learning to drive.

The long-range goal of this research is to develop a sustainable and generalizable intervention that will reduce crashes and related injuries among teen drivers by increasing safe driving practices. The investigators propose to conduct a randomized trial of an educational intervention for parents of newly licensed adolescent drivers to increase parental involvement in teaching driving skills and safe driving behavior. Seven schools in small towns in the state of Iowa have agreed to participate. These schools are all within 50 miles of Des Moines, Iowa's largest city, which will lead to driving exposure in rural and town environments.

Parents of newly-licensed teenaged drivers will be the primary subjects enrolled in this study, and parents only will participate in the intervention. Teen drivers will also be enrolled so that they can provide information about their driving attitudes and behaviors; their role will be limited to filling out surveys. The intervention will include a focus on teaching driving skills and behaviors and on effective communication strategies with teens. The intervention content includes specific driving goals that parents meet with their teen drivers that focus on skills and behavior. This project will be conducted in a rural population, so skills for driving on rural roads will be included. The delivery of the intervention will use motivational interviewing, a successful and age-appropriate health behavior communication technique that has shown great success in related health fields.

250 parent/teen dyads will be individually randomized into intervention and control groups. The intervention group will receive a tailored, in-person intervention with a trained member of the research team, with follow-up intervention phone calls each month for the 3-month intervention. The control group will be a "usual care" group who will receive driving safety materials available to all new drivers and their parents. Parents and teens will be followed to see if intervention parents meet the intervention's driving goals and to see if the parent and teens report improved driving skills and behaviors in the intervention compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* parent and teen dyads of newly-licensed teenaged drivers that speak English

Exclusion Criteria:

* siblings of previously enrolled dyads, teens who will not drive independently after licensure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Driving Safety Communication | 6 months post-intervention
Risky Driving Inventory | 6-months post intervention

SECONDARY OUTCOMES:
Driving citations and crashes | through one year post-intervention
parent risky driving inventory | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Peek-Asa, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa

REFERENCES:
- [Derived] Peek-Asa C, Cavanaugh JE, Yang J, Chande V, Young T, Ramirez M. Steering teens safe: a randomized trial of a parent-based intervention to improve safe teen driving. BMC Public Health. 2014 Jul 31;14:777. doi: 10.1186/1471-2458-14-777. PMID 25082132